CLINICAL TRIAL: NCT03222622
Title: A Multicenter, Randomized, Double-blind, Four-Arm Parallel-Group, Placebo-Controlled Phase II Study to Evaluate the Efficacy and Safety of Icotinib Hydrochloride Cream in Patients With Mild to Moderate Psoriasis
Brief Title: Study of Icotinib Hydrochloride Cream in Patients With Mild to Moderate Psoriasis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The efficacy failed to meet the primary efficacy endpoint
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Collaborators: Tigermed Consulting Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTP-16322
Record Dates: First submitted 2017-07-14; First posted 2017-07-19 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Mild to Moderate Psoriasis
Keywords: EGFR inhibitor, topical agent, psoriasis, phase 2
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): 65 patients with mild to moderate psoriasis will be randomized to receive 1% Icotinib hydrochloride cream, applied twice daily for 12 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Icotinib hydrochloride cream
- Cohort 2 (Experimental): 65 patients with mild to moderate psoriasis will be randomized to receive 2% Icotinib hydrochloride cream, applied twice daily for 12 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Icotinib hydrochloride cream
- Cohort 3 (Experimental): 65 patients with mild to moderate psoriasis will be randomized to receive 4% Icotinib hydrochloride cream, applied twice daily for 12 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Icotinib hydrochloride cream
- Cohort 4 (Placebo Comparator): 65 patients with mild to moderate psoriasis will be randomized to receive placebo cream (blank cream containing no icotinib hydrochloride), applied twice daily for 12 consecutive weeks. The drug will be applied topically to the psoriasis site.
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Icotinib hydrochloride cream — Apply topically twice daily for 12 consecutive weeks
  Other Names: no other name
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: Placebo cream — Apply topically twice daily for 12 consecutive weeks
  Other Names: no other name
  Arms: Cohort 4

SUMMARY:
This is a phase II study to evaluate the efficacy and safety of Icotinib Hydrochloride Cream in patients with mild to moderate psoriasis.

DETAILED DESCRIPTION:
Icotinib Hydrochloride is an oral, small-molecule epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor, which has been approved for treating advanced non-small cell lung cancer (NSCLC) in China. Over-expressions of EGFR and its downstream signaling proteins are implicated in the pathogenesis of psoriasis and TKIs have been considered as potential antipsoriatic agents. Icotinib hydrochloride is being developed as a cream for the treatment of mild to moderate psoriasis. This is a multicenter , randomized, doubleblind, four-arm parallel-group, placebo-controlled phase II study to assess the efficacy and safety of icotinib hydrochloride cream (1.0%, 2.0%, 4.0%) in patients with mild to moderate psoriasis. Approximately 260 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed plaque psoriasis for at least six months with multiple treatable areas (i.e. the lesion should not only on the face, scalp, genitals or skinfolds) which covers less than 10% of the total Body Surface Area (BSA), and affected area on the limb and/or trunk ≥ 1% BSA. The long diameter and thickness of target plaque psoriasis was ≥ 2cm and ≥2, respectively.
* In good health condition, with no history of diseases of major organs and no abnormality found on physical examination and vital signs.
* Men and women of childbearing potential must agree to use a contraceptive regimen agreed by the doctor during the trial. Female subjects that are on hormonal contraceptives must continue using the same hormonal contraceptive as that was used in the past 3 months, with the same route of administration and the same dose during the whole study.
* Have signed a written informed consent before entering the study.

Exclusion Criteria:

* Psoriasis guttata, psoriasis punctata, erythrodermic psoriasis, pustular psoriasis, psoriasis arthritis.
* Evidence of skin conditions other than psoriasis that would interfere with evaluations of the effect of study medication on psoriasis.
* Drug-induced psoriasis.
* Present with or had historical interstitial lung disease.
* In the opinion of the investigator, the subjects were not considered appropriate candidates.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving a 50% improvement from baseline in psoriasis area and severity index (PASI 50) score at week 8 | 8 weeks
  PASI: Combined assessment of lesion area and severity affected into single score. The body was divided into four sections [head (10% of a person's total skin); arms (20%); trunk (30%); legs (40%)]. For each section, the area of skin involved was scored from 0 (0%) to 6 (90-100%), and the severity of skin involved was estimated by clinical signs (erythema, induration, and desquamation) to score from 0 (none) to 4 (maximum). Final PASI = Sum of severity score for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 50 represents the percentage (or number) of patients who have achieved a 50% or more reduction in their PASI score from baseline.

SECONDARY OUTCOMES:
PASI 50 score at each visit through week 12 (except week 8) | Baseline to week 12 (except week 8)
  PASI: Combined assessment of lesion area and severity affected into single score. The body was divided into four sections [head (10% of a person's total skin); arms (20%); trunk (30%); legs (40%)]. For each section, the area of skin involved was scored from 0 (0%) to 6 (90-100%), and the severity of skin involved was estimated by clinical signs (erythema, induration, and desquamation) to score from 0 (none) to 4 (maximum). Final PASI = Sum of severity score for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 50 represents the percentage (or number) of patients who have achieved a 50% or more reduction in their PASI score from baseline.
Percentage of participants achieving a 75% improvement from baseline in psoriasis area and severity index (PASI 75) score at each visit through week 12 | Baseline to week 12
  PASI: Combined assessment of lesion area and severity affected into single score. The body was divided into four sections [head (10% of a person's total skin); arms (20%); trunk (30%); legs (40%)]. For each section, the area of skin involved was scored from 0 (0%) to 6 (90-100%), and the severity of skin involved was estimated by clinical signs (erythema, induration, and desquamation) to score from 0 (none) to 4 (maximum). Final PASI = Sum of severity score for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4). PASI 75 represents the percentage (or number) of patients who have achieved a 75% or more reduction in their PASI score from baseline.
Change PASI score at each visit from baseline through week 12 | Baseline to week 12
  PASI: Combined assessment of lesion area and severity affected into single score. The body was divided into four sections [head (10% of a person's total skin); arms (20%); trunk (30%); legs (40%)]. For each section, the area of skin involved was scored from 0 (0%) to 6 (90-100%), and the severity of skin involved was estimated by clinical signs (erythema, induration, and desquamation) to score from 0 (none) to 4 (maximum). Final PASI = Sum of severity score for each section * area score * weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4).
Percentage of participants achieving the physician global assessment (PGA) of psoriasis responses of clear (0) or almost clear (1) and ≥2 grade improvement at each visit through week 12 | Baseline to week 12
  PGA of Psoriasis: score based on dermatologist's assessment of skin disease averaged over all lesions. Overall lesions were graded for induration, erythema, and scaling; range: 0 (no evidence) to 5 (severe). Higher scores indicate greater severity of disease.
Lesion severity | Baseline to week 12
  Lesion severity includes the sum of 3 indications, e.g. Erythema, scaling, thickness of target psoriasis site on patients with mild to moderate psoriasis. Each indication is scored from 0 (not at all serious) to 4 (very serious).

OTHER OUTCOMES:
Safety in patients with mild to moderate psoriasis: Incidence and severity of Adverse Events, Physical Examinations, Vital signs, clinical laboratory assessments, ECG | Baseline to week 12
  Incidence and severity of Adverse Events, Physical Examinations, Vital signs (temperature, Heart Rate, blood pressure and respiration rate), clinical laboratory assessments (serum chemistry, hematology, C-reactive protein, fecal and urinalysis), ECG, etc.
Dermatology Life Quality Index (DLQI) | Baseline to week 12
  DLQI assessment includes 10 items, which encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships and side-effects of the treatment. Each item is scored from 0 (not at all relevant) to 1 (a little relevant), 2 (a lot relevant) and 3 (very much relevant). The scores of items 1-10 for change from baseline are summarized here.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zheng, PHD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No